CLINICAL TRIAL: NCT04352985
Title: Evaluating the Use of Polymyxin B Cartridge Hemoperfusion for Patients With Septic Shock and COVID 19
Status: No longer available | Type: Expanded Access
Sponsor: Spectral Diagnostics (US) Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SDI-PMX-013
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Septic Shock; Endotoxemia; COVID; Corona Virus Infection; Sepsis, Severe
MeSH Terms: conditions — Shock, Septic; Endotoxemia; Coronavirus Infections; Sepsis

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Device: Toraymyxin PMX-20R (PMX Cartridge) — The intervention is two (2) treatment sessions of PMX cartridge administration within approximately 24 hours of each other. Each treatment session will target 2 hours with a minimum of 1 ½ hours, at a flow rate of approximately 100 mL/minute, (range of 80 to 120 mL/minute). In cases where the clinical status of the subject is improving, or if the subject suffers from a relapse and the treating physician believes an additional PMX treatment may improve the clinical outcome of the subject, they may administer an additional PMX treatment session (for a total of 3 treatment sessions) at their discretion. All subjects will continue to receive standard medical care for COVID 19 and septic shock.

SUMMARY:
Prospective, observational, clinical investigation of PMX cartridge use in COVID 19 patients with septic shock

DETAILED DESCRIPTION:
This is a compassionate use protocol for a population of patients with an immediately life-threatening condition, for whom no comparable alternative therapy options are available. The PMX cartridge will be utilized to treat critically ill patients with septic shock who also have COVID 19 virus. The objective will be to observe the efficacy of the PMX cartridge with a focus on safety of use in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age
2. Hypotension requiring vasopressor support: Requirement for at least one of the vasopressors listed below, at the dose shown below, for at least 2 continuous hours and no more than 30 hours

   1. Norepinephrine > 0.05mcg/kg/min
   2. Dopamine > 10 mcg/kg/min
   3. Phenylephrine > 0.4 mcg/kg/min
   4. Epinephrine > 0.05 mcg/kg/min
   5. Vasopressin > 0.03 units/min
   6. Vasopressin (any dose) in combination with another vasopressor listed above
3. The subject must have received intravenous fluid resuscitation of a minimum of 30mL/kg administered within 24 hours of eligibility
4. Documented or suspected infection defined as definitive or empiric intravenous antibiotic administration
5. The subject must have a screening multi-organ dysfunction score (MODS) >9
6. Endotoxin Activity Assay between ≥ 0.60 to <0.90 EA units
7. Evidence of at least 1 of the following criteria for new onset organ dysfunction that is considered to be due to the acute illness:

   1. Requirement for positive pressure ventilation via an endotracheal tube or tracheostomy tube
   2. Thrombocytopenia defined as acute onset of platelet count <150,000µ/L or a reduction of 50% from prior known levels
   3. Acute oliguria defined as urine output <0.5mL/kg/hr for at least 6 hours despite adequate fluid resuscitation
8. Positive COVID 19 diagnosis

Exclusion Criteria:

1. Inability to obtain an informed consent from the subject, family member or an authorized surrogate
2. Lack of commitment for full medical support
3. Inability to achieve or maintain a minimum mean arterial pressure (MAP) of ≥ 65mmHg despite vasopressor therapy and fluid resuscitation
4. Subject has end-stage renal disease and requires chronic dialysis
5. There is clinical support for non-septic shock such as:

   1. Acute pulmonary embolus
   2. Transfusion reaction
   3. Severe congestive heart failure (e.g. NYHA Class IV, ejection fraction < 35%)
6. Subject has had chest compressions as part of CPR during this hospitalization without immediate return to communicative state
7. Subject has had an acute myocardial infarction (AMI) within the past 4 weeks
8. Subject has uncontrolled hemorrhage (acute blood loss requiring > 3 UPC in the past 24 hours)
9. Major trauma within 36 hours of screening
10. Subject has severe granulocytopenia (leukocyte count less than 500 cells/mm3) or severe thrombocytopenia (platelet count less than 30,000 cells/mm3)
11. HIV infection in association with a last known or suspected CD4 count of <50/mm3
12. Subject's baseline state is non-communicative
13. Subject has sustained extensive third-degree burns within the past 7 days
14. Body weight < 35 kg (77 pounds)
15. Known hypersensitivity to Polymyxin B
16. Subject has known sensitivity or allergy to heparin or has a history of heparin associated thrombocytopenia (H.I.T.)
17. Subject is currently enrolled in an investigational drug or device trial
18. Subject has been previously enrolled in the current trial
19. Any other condition, that in the opinion of the investigator, would preclude the subject from being a suitable candidate for enrollment, such as end-stage chronic illness (eg. lack of source control and bowel necrosis) with no reasonable expectation of survival to hospital discharge

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Connecticut Health Center, Farmington, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Stony Brook University Hospital, Stony Brook, New York